CLINICAL TRIAL: NCT02237820
Title: Dexamethasone Versus Prednisone in Heart Failure Patients, Hospitalized With Exacerbation of Chronic Obstructive Pulmonary Disease.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Gideon Stein, md, MD , PhD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: no specific protocol ID
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — Dexamethasone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone
- Prednisone (Active Comparator)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Dexamethasone — 6 mg/day of Oral Dexamethasone
  Arms: Dexamethasone
Drug: Prednisone — 40 mg/day of Oral Prednisone
  Arms: Prednisone

SUMMARY:
This is the first study assessing the impact of dexamethasone (a glucocorticosteroid with negligible mineralocorticoid activity) as compared to prednisone on short-term outcomes of HF patients hospitalized with exacerbation of COPD. The study may provide important data regarding a simple but potentially robust intervention among large patient population with high rates of hospital admissions.

DETAILED DESCRIPTION:
An Open-label randomized prospective study of HF patients (NYHA grade II-VI), hospitalized with COPD exacerbation. Eighty patients will be randomized in a 1:1 fashion to conventional and intervention testament groups. Informed consent will be obtained from all patients prior to study enrolment.

Randomization will be performed using RED cap - secure web application. The conventional therapy group will receive 40mg of oral prednisone daily, while the intervention group will be treated with oral dexamethasone in an equivalent anti-inflammatory dose of 6 mg/day. Glucocorticosteroids will be administered throughout hospitalization and will be continued for at least 5-7 days. Dose changes through this period, as well as subsequent tapering will be on the discretion of the treating physician. All patients will also be treated with short-acting bronchodilators, antibiotics, oxygen, positive pressure non-invasive mechanical ventilation and VTE prophylaxis - based on the GOLD 2019 guidelines and clinical judgment of the attending physicians. An order for low sodium diet will be written. Discharge decisions will be based on the GOLD 2019 discharge criteria list. Patients will be discharge without steroid tapering regimen unless indicated by clinical judgment. Patient's demographic data will be documented at baseline (age, sex, GOLD severity stage, data on hospitalizations in the past year, patients' chronic drug therapy, Last spirometry and two-dimensional echo-Doppler examination results).

On admission, patients' weight, height and oxygen saturation will be measured and routine blood tests will be drawn for evaluation of complete blood count, chemistry, NT proBNP levels, troponin, C-reactive protein and venous blood gas. Blood test results will be taken from the patient electronic medical record and will be based on the tests taken in the ER and during ward admission. Upon recruitment, the patient will be asked to complete COPD assessment tool (CAT) questionnaire and the Kansas City Cardiomyopathy Questionnaire (KCCQ-12, the short form version) in order to quantify their health status. A follow-up telephone call visit will be performed 14±2 and 28±2 days after enrollment. The following measures will be obtained: KCCQ-12 and CAT questionnaire scores and documentation of current diuretic dose. After study completion, each patient will be followed for 30 more days post admission in order to document further hospitalizations.

All the date collected during the study and after patients enrollment will be documented on a specialized case report form (CRF) built on RED cap - secure web application.

ELIGIBILITY:
Inclusion criteria:

* Age > 40 years.
* Patients with a previous diagnosis of COPD and evidence of airflow limitation (GOLD severity stage of II-IV).
* Patients with COPD exacerbation and potential indications for hospitalization as defined by the 2019 GOLD guidelines.
* Patients with a diagnosis of heart failure (NYHA grade II-IV).

Exclusion criteria:

* Patients with a severe exacerbation on enrollment, based upon arterial PH<7.2 or PaCO2 > 90 mmHg
* Patients who are currently participating in other studies.
* Known hypersensitivity to prednisone / dexamethasone.
* Patients who were treated with systemic corticosteroids one month prior to admission, unless prednisone dosage is 20 mg or less.
* Patients who are unable to provide an informed consent.
* Pregnant woman.
* Patients on Chronic mechanical ventilation.

Study drug treatment termination criteria:

* Hypersensitivity reaction to prednisone / dexamethasone.
* Any clinical deterioration, which at the discretion of the treating physician and/or study investigators, necessitate change of the study steroid treatment (such as, but not limited to, need to stop oral medication).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | up to 1 month
Change in COPD assessment tool (CAT) questionnaire score | Baseline, Week 2, Week 4
Change in the Kansas City Cardiomyopathy Questionnaire (KCCQ-12 short form) score | Baseline, Week 2, Week 4

SECONDARY OUTCOMES:
Rate of re-admission | 30 days post enrollment
  rate of respiratory deterioration necessitate intubation, re-admission or death at 30-day post enrollment

OTHER OUTCOMES:
Change from Baseline in diuretic doses | Baseline, Week 2, Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Y Stein, MD PhD, Principal Investigator — Beilinson Hospital, Rabin Medical Center; Ran Nissan, PharmD, Study Director — Beilinson Hospital, Rabin Medical Center; Lisa Cooper, MD, Study Director — Beilinson Hospital, Rabin Medical Center; Mordechai R Kramer, MD, Principal Investigator — Beilinson Hospital, Rabin Medical Center; Shmuel Fuchs, MD, Principal Investigator — Beilinson Hospital, Rabin Medical Center
Locations (1):
- Beilinson Hospital, Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Hawkins NM, Petrie MC, Jhund PS, Chalmers GW, Dunn FG, McMurray JJ. Heart failure and chronic obstructive pulmonary disease: diagnostic pitfalls and epidemiology. Eur J Heart Fail. 2009 Feb;11(2):130-9. doi: 10.1093/eurjhf/hfn013. PMID 19168510
- [Background] Iversen KK, Kjaergaard J, Akkan D, Kober L, Torp-Pedersen C, Hassager C, Vestbo J, Kjoller E; ECHOS-Lung Function Study Group. Chronic obstructive pulmonary disease in patients admitted with heart failure. J Intern Med. 2008 Oct;264(4):361-9. doi: 10.1111/j.1365-2796.2008.01975.x. Epub 2008 Jun 5. PMID 18537871
- [Background] Iversen KK, Kjaergaard J, Akkan D, Kober L, Torp-Pedersen C, Hassager C, Vestbo J, Kjoller E; ECHOS Lung Function Study Group. The prognostic importance of lung function in patients admitted with heart failure. Eur J Heart Fail. 2010 Jul;12(7):685-91. doi: 10.1093/eurjhf/hfq050. Epub 2010 Apr 15. PMID 20395261
- [Background] Schweiger TA, Zdanowicz M. Systemic corticosteroids in the treatment of acute exacerbations of chronic obstructive pulmonary disease. Am J Health Syst Pharm. 2010 Jul 1;67(13):1061-9. doi: 10.2146/ajhp090293. PMID 20554591
- [Background] Maxwell CB, Jenkins AT. Drug-induced heart failure. Am J Health Syst Pharm. 2011 Oct 1;68(19):1791-804. doi: 10.2146/ajhp100637. PMID 21930637
- [Background] Wei L, MacDonald TM, Walker BR. Taking glucocorticoids by prescription is associated with subsequent cardiovascular disease. Ann Intern Med. 2004 Nov 16;141(10):764-70. doi: 10.7326/0003-4819-141-10-200411160-00007. PMID 15545676
- [Background] Global Initiative for Chronic Obstructive Lung Disease (GOLD). Updated 2013.
- [Background] Gardner D, Shoback D. Greenspan's basic & clinical endocrinology, 9 edition. McGraw-Hill Companies, Inc.